CLINICAL TRIAL: NCT00140543
Title: A European Multicenter Open-Label Randomised Trial to Evaluate the Efficacy and Safety of Sirolimus and Tacrolimus Compared to MMF and Tacrolimus With Short-Course Induction Therapy, Short-Term Steroids Application in de Novo SPK Transplanted Diabetic Patients
Brief Title: European Trial of Immunosuppression in SPK Tx
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EUROSPK Study Group (Other)
Collaborators: Fujisawa GmbH (Industry); Hoffmann-La Roche (Industry); Wyeth is now a wholly owned subsidiary of Pfizer (Industry); Neovii Biotech (Industry); Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUROSPK002
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus, Type 1; Diabetic Nephropathy
Keywords: simultaneous pancreas/kidney transplantation; Immunosuppression
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Nephropathies

INTERVENTIONS:
Drug: sirolimus versus mycophenolate mofetil

SUMMARY:
1. To determine and compare the efficacy of Tacrolimus/Rapa versus Tacrolimus/MMF-based immunosuppression (in conjunction with initial short-term steroids and polyclonal antibody administration) in Type 1-diabetic patients undergoing simultaneous pancreas/kidney allograft transplantation.
2. To evaluate the safety of Tacrolimus/Rapa versus Tacrolimus/MMF in terms of drug-related complications and overimmunosuppression-associated complications, particularly under monitoring of the pharmacokinetic profile of all drugs administered.

DETAILED DESCRIPTION:
This will be a controlled, randomised study, to be performed in 15-20 pancreas transplantation centers throughout Europe. Patients will be randomised into one of two treatment groups. Group 1 will receive Tacrolimus and Mycophenolate Mofetil (= best group in EuroSPK001 trial). Group 2 will receive Tacrolimus and Sirolimus. Both groups will receive in association short-term corticosteroids and polyclonal antibody preparation. Patients will be randomly assigned to one of the 2 treatment groups in a 1:1 ratio before transplantation. The study will last 3 years, with a first interim analysis of the data at 6 months and a complete analysis at 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, of 18 to 55 years of age, with end-stage, C-peptide-negative, Type 1-diabetic nephropathy.
2. Female patients of childbearing age must have a negative pregnancy test and must agree to maintain effective birth control practice throughout the study period (3 years).
3. Patient must have signed the Patient Informed Consent Form.
4. Patient must receive a primary simultaneous pancreas/kidney (SPK) cadaveric transplant, with either intestinal or bladder and either portal or systemic venous drainages.

Exclusion Criteria:

1. Patient is pregnant or breastfeeding.
2. Patient is allergic or intolerant to Mycophenolate Mofetil, Sirolimus, Tacrolimus or other macrolides, or any compounds structurally related to these compounds.
3. Patient has a positive T-cell crossmatch on the most recent serum specimen.
4. Patient is known for active liver disease or has significant liver disease, defined by ASAT and ALAT serum levels greater than 3 times the upper limit of normal.
5. Patient has malignancy or history of malignancy, with the exception of adequately treated localised squamous cell or basal cell carcinoma, without recurrence.
6. Patient has been included in another clinical trial protocol for any investigational drug within 4 weeks prior to randomisation.
7. Patient has any form of substance abuse, psychiatric disorder or condition, which, in the opinion of the investigator, may invalidate communication.
8. Patient receives a SPK transplant from a living donor, or receives segmental pancreatic transplant, or a previous kidney transplant alone.
9. Pancreatic duct occlusion technique .
10. Donor is older than 55 years of age.

    -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 228
Dates: Start 2002-02; Study Completion 2005-09-30 (Actual)

PRIMARY OUTCOMES:
At 1 year:Incidence of biopsy-proven (kidney) rejection episodes.

SECONDARY OUTCOMES:
SECONDARY ENDPOINTS: At 6 months and 1 year
* Kidney/Pancreas function (at 6 months and 1 year):
- Kidney function will be measured by:
- S- creatinine
- Creatinine clearance
- Pancreas function will be measured by:
- Fasting Glucose level (< 123 mg/dl)
- HbA1C
- Need for insulin therapy
- Need for oral drugs
* At 6 months and 1 year:
- Patient and graft survival
- Lipid profile
- Infections
- Side effects
- Blood Pressure
- Treatment failure for any reason, such as permanent discontinuation of a drug, graft loss or death.
* % of steroid free patients: at 6 months and 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Squifflet, MD,PhD, Study Chair — SPEAKER FOR THE EUROSPK STUDY GROUP
Locations (14):
- Universitätsklinik, Innsbruck, Austria
- Belgium (3):
  - Cliniques Universitaires Saint Luc, Brussels
  - UZ Gent, Ghent
  - UZ Gasthuisberg, Leuven
- Institute for clinical and experimental medicine-IKEM, Prague, Czechia
- Germany (6):
  - Charite Campus Virchow Klinikum, Berlin
  - Goethe University, Frankfurt am Main
  - Chirurgische Universitätsklinik, Freiburg im Breisgau
  - Knappschaftskrankenhaus, Langendreer
  - Klinikum Grosshadern-University of Munich, Munich
  - Klinikum Innenstadt der Universität München, Munich
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Hospital Clinico, Barcelona, Spain
- Hôpital Cantonal de Geneve, Geneva, Switzerland